CLINICAL TRIAL: NCT05392699
Title: An Open-blind Dose Escalation Study to Assess the Safety, Tolerability, and Preliminary Efficacy of ABOD2011 in Patients With Advanced Solid Tumors Progressed After Standard Systemic Therapy
Brief Title: ABOD2011 in Patients With Advanced Solid Tumors Progressed After Standard Systemic Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABOD2011-001
Record Dates: First submitted 2022-03-15; First posted 2022-05-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human single chain IL-12 mRNA-single dose (Experimental): Human single chain IL-12 mRNA-single dose
  Interventions: Biological: human single chain IL-12 mRNA-single dose
- Human single chain IL-12 mRNA-multiple dose (Experimental): Human single chain IL-12 mRNA-multiple dose
  Interventions: Biological: human single chain IL-12 mRNA-multiple dose

INTERVENTIONS:
Biological: human single chain IL-12 mRNA-single dose — human single chain IL-12 mRNA administered as specified in the treatment arm with injection once only
  Arms: Human single chain IL-12 mRNA-single dose
Biological: human single chain IL-12 mRNA-multiple dose — human single chain IL-12 mRNA administered as specified in the treatment arm with injection once per week for 3 weeks
  Arms: Human single chain IL-12 mRNA-multiple dose

SUMMARY:
Based on the activation and regulation of immune system by cytokines, mRNA encoding cytokines has become one of the important directions of mRNA tumor drug development. This product (ABOD2011) is a new generation mRNA product for intratumoral injection.

The primary objective of this study is to assess the safety and tolerability, of ABOD2011 in patients with advanced solid tumors that progressed after standard systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older.
2. Understand and voluntarily sign the informed consent form (ICF).
3. Histopathologically confirmed recurrent or metastatic solid tumors.
4. Failure of prior systemic standard of care, or intolerance to severe toxicity, or lack of standard of care.
5. Presence of at least one measurable lesion as assessed by RECIST Version 1.1.
6. At least one superficial or deep lesion for intratumoral administration and biopsy.
7. Sufficient organ functions.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
9. Weight > 30 kg.
10. Expected survival longer than 12 weeks.
11. Evidence of menopause in female patients, or for women of childbearing potential: negative for urine or blood pregnancy.

Exclusion Criteria:

1. Any systemic anti-tumor therapy, within 28 days prior to the first dose.
2. Radiotherapy within 14 days prior to first dose.
3. Use of immunosuppressants.
4. Major surgery within 28 days.
5. Inadequately controlled diseases.
6. Active autoimmune and inflammatory diseases.
7. Clinically symptomatic central nervous system tumors or metastases.
8. Toxicity of prior anti-tumor therapy is still NCI-CTCAE ≥ 2.
9. Other malignancies within the previous 5 years with the exception of cured basal cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the breast, and carcinoma in situ of the cervix.
10. Active infections.
11. Other conditions that may increase the risk associated with the study drug, or affect the study compliance, etc., which, in the opinion of the investigator, are not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing dose-limiting toxicities (DLTs) | From first dose to Day 28
  Number of Participants Experiencing dose-limiting toxicities (DLTs)
Number of Participants Experiencing Adverse Events (AEs) | From signed ICF until the date of last visit or start new antitumor therapy, whichever comes first, assessed up to 36 months
  Number of Participants Experiencing Adverse Events (AEs)
Number of Participants Experiencing Severe Adverse Events (SAEs) | From signed ICF until the date of last visit or start new antitumor therapy, whichever came first, assessed up to 24 months
  Number of Participants Experiencing Severe Adverse Events (SAEs)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 36 months
  Overall Response Rate (ORR)
Disease Control Rate(DCR) | Up to 36 months
  Disease Control Rate(DCR)
Duration of Response (DOR) | Up to 36 months
  Duration of Response (DOR)
Progression-Free Survival (PFS) | Up to 36 months
  Progression-Free Survival (PFS)
Overall Survival | Up to 36 months
  Overall Survival
Maximum observed concentration (Cmax) of ABOD2011 | From first dose of ABOD2011 through to 28 days after last dose of investigational product
  Maximum observed concentration (Cmax) of ABOD2011
Area under the concentration-time curve (AUC) of ABOD2011 | From first dose of ABOD2011 through to 28 days after last dose of investigational product
  Area under the concentration-time curve (AUC) of ABOD2011
Maximum observed concentration (Cmax) of IL-12 | From first dose of ABOD2011 through to 28 days after last dose of investigational product
  Maximum observed concentration (Cmax) of IL-12
Area under the concentration-time curve (AUC) of IL-12 | From first dose of ABOD2011 through to 28 days after last dose of investigational product.
  Area under the concentration-time curve (AUC) of IL-12
Plasma concentration of IFN gamma | From first dose of ABOD2011 through to 28 days after last dose of investigational product.
  Plasma concentration of IFN gamma

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China